CLINICAL TRIAL: NCT00677183
Title: Development of a Biomarker for Development of Non-Alcoholic Steatohepatitis (NASH) in Children
Brief Title: Development of Biomarker for Development of Non-Alcoholic Steatohepatitis (NASH) in Children
Acronym: NASH
Status: Withdrawn | Type: Observational
Why Stopped: PI did not receive funding for this PI-initiated study. PI subsequently left the institution.
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Other Study IDs: CHW 08/36; GC 618
Record Dates: First submitted 2008-05-09; First posted 2008-05-14 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Non-Alcoholic Steatohepatitis
Keywords: NASH; Biomarker
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 10mL of blood will be retained from each participant and their parents. 5mL of this blood will undergo DNA extraction and genotyping for several known NASH related genes. The other 5mL of blood will be saved as serum for future analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SN###.#1: All children in this cohort will have biopsy-proven NASH.
- SN###.#2: This cohort will be parents (mother and father when possible) of child subjects with biopsy-proven NASH.

SUMMARY:
The purpose of this study is to document how often specific genotypes known to be associated with adult-onset NASH (Non-Alcoholic Steatohepatitis) occur in a pediatric cohort and investigate whether these genotypes are associated with increased susceptibility to NASH.

DETAILED DESCRIPTION:
NASH is a clinico-pathological entity characterized by the development of histological changes of inflammation and fibrosis in the liver that are nearly identical to those induced by excessive alcohol intake, but in the absence of alcohol abuse. Nonalcoholic steatohepatitis occurs commonly children with additional comorbidities such as obesity and diabetes mellitus. Paralleling the increasing prevalence of obesity and type 2 diabetes in the pediatric population, nonalcoholic fatty liver disease (NAFLD) and especially its more severe histological form NASH, is expected to become one of the most common causes of end-stage liver disease in both children and young adults.

Although no genome wide association studies have been conducted in association with NASH to date, individual candidate gene investigations have identified several genes associated with increase susceptibility to NASH in adults including the microsomal triglyceride transfer protein (MTP) which regulates the incorporation of triglycerides into apolipoprotein B and a key enzyme for the assembly and secretion of VLDL from hepatocytes, the manganese superoxide dismutase (MnSOD) gene which catalyzes the conversion of two molecules of superoxide anion, a highly unstable ROS, into hydrogen peroxide and oxygen more stable ROS, and lastly, phosphatidylethanolamine N-methyltransferase (PEMT) which is required for hepatic secretion of triacylglycerol in very low density lipoproteins (VLDL).

We propose the following aim:

Aim 1: To document the frequency of specific genotypes, previously identified to be associated with adult-onset NASH, in a purely pediatric cohort.

Aim 2: To investigate whether these genotypes are associated with increased susceptibility to NASH and increased occurrence of fibrosis in the cohort of pediatric subjects. Our hypothesis would be:

A significantly higher proportion of the polymorphisms would exist in those subjects with NASH compared to controls.

Aim 3: To investigate the presence of other polymorphisms or other biomarker that are indicative of pediatric NASH. Such that our secondary hypothesis would be:

Specific polymorphisms or biomarkers will be identified that will indicate a higher probability of NASH.

ELIGIBILITY:
Inclusion Criteria:

* All subjects aged 2-18 with biopsy proven NAFLD and/or NASH undergoing a blood draw and willing to consent to this study will qualify for inclusion in this protocol.

Exclusion Criteria:

* other causes of chronic liver disease or other chronic diseases, specifically autoimmune disorders, immunodeficiencies, or individuals with congenital/genetic disorders
* chronic viral hepatitis, Wilson's disease, or alpha -1- antitrypsin deficiency
* acute life threatening illness or conditions

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The child subjects will be recruited from the Hepatology Clinic at Children's Hospital of Wisconsin.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
We will compare known frequencies from the Hapmap and specifically compare the proportions for those with NASH in adults to see if there is a difference in the child incidence of NASH. | three years
We will compare the proportions of those with NASH to those without NASH and those with fibrosis compared to those without fibrosis. | Three years

CONTACTS AND LOCATIONS:
Overall Officials: Vincent F Biank, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Angulo P, Keach JC, Batts KP, Lindor KD. Independent predictors of liver fibrosis in patients with nonalcoholic steatohepatitis. Hepatology. 1999 Dec;30(6):1356-62. doi: 10.1002/hep.510300604. PMID 10573511
- [Background] Huang BE, Amos CI, Lin DY. Detecting haplotype effects in genomewide association studies. Genet Epidemiol. 2007 Dec;31(8):803-12. doi: 10.1002/gepi.20242. PMID 17549762
- [Background] Benjamini, Y. and Hochberg, Y. 1995. Controlling the false discovery rate: A practical and powerful approach to multiple testing. J. Royal Stat. Soc. B (57): 289-300.
- [Background] Breiman L, Friedman JH, Olshen RA, Stone CJ. Classification and Regression Trees. Classification and Regression Trees. 1984.
- [Background] Lin DY, Zeng D, Millikan R. Maximum likelihood estimation of haplotype effects and haplotype-environment interactions in association studies. Genet Epidemiol. 2005 Dec;29(4):299-312. doi: 10.1002/gepi.20098. PMID 16240443
- [Background] Iacobellis A, Marcellini M, Andriulli A, Perri F, Leandro G, Devito R, Nobili V. Non invasive evaluation of liver fibrosis in paediatric patients with nonalcoholic steatohepatitis. World J Gastroenterol. 2006 Dec 28;12(48):7821-5. doi: 10.3748/wjg.v12.i48.7821. PMID 17203527
- [Background] Marra F. NASH: are genes blowing the hits? J Hepatol. 2004 May;40(5):853-6. doi: 10.1016/j.jhep.2004.03.005. No abstract available. PMID 15094235
- [Background] Song J, da Costa KA, Fischer LM, Kohlmeier M, Kwock L, Wang S, Zeisel SH. Polymorphism of the PEMT gene and susceptibility to nonalcoholic fatty liver disease (NAFLD). FASEB J. 2005 Aug;19(10):1266-71. doi: 10.1096/fj.04-3580com. PMID 16051693
- [Background] Marshall RJ. Partitioning methods for classification and decision making in medicine. Stat Med. 1986 Sep-Oct;5(5):517-26. doi: 10.1002/sim.4780050516. PMID 3538265